CLINICAL TRIAL: NCT01466569
Title: A Phase 1 A/B Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AbGn-7 Therapy Alone and in Combination With the FOLFOX7 Treatment Regimen in Patients With Advanced Solid Tumors
Brief Title: An A/B Dose Escalation Study of AbGn-7 Alone and With FOLFOX7 Treatment in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbGenomics B.V Taiwan Branch (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AbGenomics-2010.007.01
Record Dates: First submitted 2011-11-02; First posted 2011-11-08 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Solid Tumor of Epithelial Origin; Gastric Cancer
Keywords: Advanced Solid Tumor; Gastric Cancer; Oncology; monoclonal Antibody
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- AbGn-7 phase 1a cohort 1 (Experimental)
  Interventions: Drug: AbGn-7
- AbGn-7 phase 1a cohort 2 (Experimental)
  Interventions: Drug: AbGn-7
- AbGn-7 phase 1a cohort 3 (Experimental)
  Interventions: Drug: AbGn-7
- AbGn-7 phase 1b cohort 1 (Experimental)
  Interventions: Drug: AbGn-7
- AbGn-7 phase 1b cohort 2 (Experimental)
  Interventions: Drug: AbGn-7

INTERVENTIONS:
Drug: AbGn-7 — Phase 1a: dose escalation; Drug: AbGn-7 weekly iv infusion Duration: 6 weeks
  Arms: AbGn-7 phase 1a cohort 1; AbGn-7 phase 1a cohort 2; AbGn-7 phase 1a cohort 3
Drug: AbGn-7 — Phase 1b: two doses (one dose below MTD/MAD and MTD/MAD as determined in phase 1a) Drug: AbGn-7 weekly iv infusion combined with FOLFOX7 Duration: 6 weeks
  Arms: AbGn-7 phase 1b cohort 1; AbGn-7 phase 1b cohort 2

SUMMARY:
The purpose of this study is to determine the safety and tolerability profile including the dose limiting toxicity of AbGn-7 in patients with chemo-refractory advanced solid tumor of epithelial origin, and of AbGn-7 in combination with FOLFOX7 in patients with chemo-naive/chemo-refractory recurrent, locally advanced or metastatic gastric cancer.

DETAILED DESCRIPTION:
Monoclonal antibodies, alone or in combination with chemotherapeutic agents, have been proven to be effective treatment for many malignant diseases in human. Antibodies can mediate cytotoxicity through complement dependent cytotoxicty (CDC), antibody dependent cell mediated cytotoxicity (ADCC) or apoptosis.

AbGn-7 was identified based on its direct killing (apoptosis-inducing) activities towards cancer cells expressing its epitope. In vitro data also demonstrated its ability to elicit CDC and ADCC. The in vivo xenograft study of AbGn-7 demonstrated that AbGn-7 alone or in combination with chemotherapeutic agents successfully suppressed the growth of gastric, pancreatic, and colorectal tumours. The NHP study proved the safety profile of AbGn-7. The present Phase 1 clinical study is designed to evaluate the safety and tolerability of AbGn-7 alone in patients with solid tumors of epithelial origin (Phase 1a) and in combination with a current chemotherapeutic regimen FOLFOX7 in patients with recurrent, locally advanced or metastatic gastric carcinoma (Phase 1b).

ELIGIBILITY:
Inclusion Criteria:

1. must provide written informed consent.
2. must be ≥18 years of age, either sex and of any race/ethnicity.
3. Phase 1a: must have a histologically or cytologically confirmed advanced malignant solid tumor of epithelial origin and must have failed on previous chemotherapy. Phase 1b: must have a histologically or cytologically confirmed, recurrent, locally advanced or metastatic gastric cancer with measurable disease; must be chemo-naïve or must have failed on previous chemotherapy; must not have received an oxaliplatin-based chemotherapeutic regimen or monoclonal antibody therapy.
4. must have an Eastern Cooperative Oncology Group Performance Status of ≤2.
5. must have adequate hematological, renal and liver functions within 3 weeks prior to first study drug administration as evidenced by: a) Absolute neutrophil count ≥1.5 x 109/L, b) Hemoglobin ≥90 g/L (≥80 g/L for patients with documented renal cell carcinoma), c) Platelet count ≥100 x 109/L, d) Serum creatinine ≤1.5 x upper limit of normal ULN or a calculated creatinine clearance ≥60 mL/minute, e) Total bilirubin <1.5 x ULN, except for patients with documented Gilbert's disease, f) AST/SGOT and ALT/SGPT < 2.5 x ULN, or, in the presence of documented liver metastases, ≤5 x ULN.
6. must be able to adhere to dose and visit schedules.
7. Each female patient of childbearing potential must agree to use a medically accepted method of contraception or to abstain from sexual intercourse and each male patient must agree to use a medically accepted method of contraception or to abstain from sexual intercourse during the study and for 60 days after stopping the study drug.
8. A life expectancy of at least 3 months.
9. Available tumor tissue in the form of unstained slides for determination of AbGn-7 epitope expression (optional for Phase 1a, obligatory for Phase 1b). Patients without archival/banked tumor tissue obtained at the time of initial diagnosis must have a biopsy performed according to institutional guidelines prior to the initiation of treatment.

Exclusion Criteria:

1. No current treated or untreated leptomeningeal metastasis or a metastatic CNS lesion.
2. For Phase 1a, patients should not have received chemotherapy within 30 days prior to initiation of AbGn-7 therapy. For Phase 1b, patients should not have received oxaliplatin-based chemotherapy or monoclonal antibody therapy for their gastric cancer prior to enrollment.
3. Have note received radiation therapy within 3 weeks prior to first study drug administration and must have adequately recovered from any associated toxicity and/or complications of this intervention.
4. Have not undergone major surgery within 3 weeks prior to the first study drug administration and must have adequately recovered from the toxicity and/or complications of these interventions.
5. No current human immunodeficiency virus (HIV) infection or a current HIV-related malignancy.
6. No current active hepatitis B or C.
7. No any serious or uncontrolled infection.
8. No uncontrolled diabetes mellitus, defined as a HbA1c of ≥7.5% in a patient with documented diabetes mellitus.
9. No any of the following within 6 months prior to first study drug administration: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, clinically significant cardiac dysrhythmia or clinically significant ECG abnormality, cerebrovascular accident or transient ischemic attack, or seizure disorder.
10. No persistent, unresolved NCI CTCAE Grade ≥2 drug-related toxicity associated with previous chemotherapy.
11. Not participating in any other clinical study with a potentially therapeutic agent, or have not received another investigational product within 21 days.
12. No any clinically significant condition or situation which would interfere with the study evaluations or optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety will be assessed by analysis of adverse event, clinical laboratory tests and physical examination | 10 Weeks

SECONDARY OUTCOMES:
Pharmacokinetics will be assessed at 3 different dose levels in phase 1a and at 2 dose levels in phase 1b | 12 Weeks
Serum anti-drug antibodies will be assessed at 3 different dose levels in phase 1a and at 2 dose levels in phase 1b | 12 weeks
Tumor response rate by Response Evaluation Criteria in Solid Tumors (RECIST) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yao Lin, MD, PhD, Study Director — AbGenomics B.V Taiwan Branch; Devalingham Mahalingam, MD, Principal Investigator — The University of Texas Health Science Center-CTRC; Anthony Olaszanski, MD, RPh, Principal Investigator — Fox Chase Cancer Center; Kuen-Hui Yeh, MD, Principal Investigator — National Taiwan University Hospital; Ruey-Kuen Hsieh, MD, Principal Investigator — Mackay Memorial Hospital
Locations (4):
- United States (2):
  - Fox Chase Cancer Center, Rockledge, Pennsylvania
  - The University of Texas Health Science Center-CTRC, San Antonio, Texas
- Taiwan (2):
  - MacKay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei